CLINICAL TRIAL: NCT03587077
Title: Effect of Adding Vaginal Isosorbide Mononitrate to Misoprostol Prior to Intrauterine Device Insertion in Women Delivered Only by Elective Cesarean Section: a Randomized Double-blind Controlled Clinical Trial
Brief Title: Pain Relief During IUD Insertion in Women Delivered Only by Elective Cesarean Section
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Eman Ibrahim Ramadan Abdelrahman, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pain during IUD insertion
Record Dates: First submitted 2018-04-09; First posted 2018-07-16 (Actual); Last update posted 2018-07-16 (Actual); Status verified 2018-06

CONDITIONS: IUD Insertion Complication
MeSH Terms: interventions — Misoprostol; isosorbide-5-mononitrate

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): Women will receive vaginally one tablet misoprostol 200 mcg(Misotac; Sigma Pharma, SAE, EGYPT) plus one tablet isosorbide mononitrate 40 mg(Effox 40 mg; Minapharm). A trained clinical nurse will introduce the tablets, digitally without using speculum, 3 hours before IUD insertion into the posterior vaginal fornix of the woman while lying in the lithotomy position.
  Interventions: Drug: Misoprostol; Drug: isosorbide mononitrate
- control group (Placebo Comparator): Women will receive vaginally one tablet misoprostol 200 mcg Plus one tablet placebo.A trained clinical nurse will introduce the tablets, digitally without using speculum, 3 hours before IUD insertion into the posterior vaginal fornix of the woman while lying in the lithotomy position.
  Interventions: Drug: Misoprostol; Drug: Placebos

INTERVENTIONS:
Drug: Misoprostol — vaginal application
Drug: Placebos — vaginal application
  Arms: control group
Drug: isosorbide mononitrate — vaginal application
  Arms: study group

SUMMARY:
The aim of the work is to assess the effect of combined misoprostol 200 mcg and isosorbide mononitrate 40 mg versus misoprostol 200 mcg and placebo as local vaginal tablet on the successful IUD insertion.

DETAILED DESCRIPTION:
Fear of pain during insertion of an IUD may deter women from choosing the IUD as a method of contraception. According to Hubacher et al. predictors of increased pain during IUD insertion include nulliparity, age greater than 30 years, lengthier time since last pregnancy or last menses, and not currently breastfeeding. Allen et al. predicted pain to be greater based on history of no previous vaginal delivery, and difficulty of the procedure. Pharmacological interventions for pain control during IUD insertion include analgesics, local anesthetics, and the use of prostaglandins to soften the cervix; however, there is wide variation in the use of these methods . Misoprostol has also been proposed as an agent to ease IUD insertion and decrease procedure-associated pain .

Nitrous oxide has been used for years for procedural analgesia in outpatient settings and has recently been investigated as an approach to pain management in the context of IUD insertion .

Sewell and Vincent have been offering nitrous oxide for reducing the pain of IUD insertion and have had a positive response.

ELIGIBILITY:
Inclusion Criteria:We will include

* Nonpregnant women,
* aged 18-45 years, .delivered before only by elective CS and did not receive any analgesics in the 24 h prior to IUD insertion.

Exclusion Criteria:We will exclude

* Women with any uterine abnormalities as congenital anomalies,
* Women with endometrial lesions,
* Women with adenomyosis,
* Women with fibroids,
* Women with intrauterine adhesions,
* Women with chronic pelvic pain,
* Women with spasmodic dysmenorrhea,
* Women with abnormal uterine bleeding,
* Women with history of cervical surgery, .Women with allergy to misoprostol or isosorbide mononitrate or any medical disease that contraindicates its use and those who refused to participate in the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — All eligible participants included in the study signed a written informed consent before participation after explaining the nature of the study.
Enrollment: 113 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2019-04 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
rate of successful IUD insertion | 10 minutes
  Defined by a distance from the IUD to the endometrial end of less than 25 mm

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad S. Abdellah, Prof., Principal Investigator — Supervisor; Ihab M. El-Nashar, Prof., Principal Investigator — Supervisor

REFERENCES:
- [Background] Akintomide H, Sewell RD, Stephenson JM. The use of local anaesthesia for intrauterine device insertion by health professionals in the UK. J Fam Plann Reprod Health Care. 2013 Oct;39(4):276-80. doi: 10.1136/jfprhc-2012-100486. Epub 2013 Feb 5. PMID 23385310
- [Background] Allen RH, Bartz D, Grimes DA, Hubacher D, O'Brien P. Interventions for pain with intrauterine device insertion. Cochrane Database Syst Rev. 2009 Jul 8;(3):CD007373. doi: 10.1002/14651858.CD007373.pub2. PMID 19588429
- [Background] Allen RH, Carey MS, Raker C, Goyal V, Matteson K. A prospective cohort study of pain with intrauterine device insertion among women with and without vaginal deliveries. J Obstet Gynaecol. 2014 Apr;34(3):263-7. doi: 10.3109/01443615.2013.868424. Epub 2014 Jan 31. PMID 24483244
- [Background] Allen RH, Raker C, Goyal V. Higher dose cervical 2% lidocaine gel for IUD insertion: a randomized controlled trial. Contraception. 2013 Dec;88(6):730-6. doi: 10.1016/j.contraception.2013.07.009. Epub 2013 Aug 1. PMID 24012096
- [Background] Asker C, Stokes-Lampard H, Beavan J, Wilson S. What is it about intrauterine devices that women find unacceptable? Factors that make women non-users: a qualitative study. J Fam Plann Reprod Health Care. 2006 Apr;32(2):89-94. doi: 10.1783/147118906776276170. PMID 16824298
- [Background] Bahamondes L, Mansour D, Fiala C, Kaunitz AM, Gemzell-Danielsson K. Practical advice for avoidance of pain associated with insertion of intrauterine contraceptives. J Fam Plann Reprod Health Care. 2014 Jan;40(1):54-60. doi: 10.1136/jfprhc-2013-100636. Epub 2013 Sep 27. PMID 24076534
- [Background] Barber EL, Lundsberg LS, Belanger K, Pettker CM, Funai EF, Illuzzi JL. Indications contributing to the increasing cesarean delivery rate. Obstet Gynecol. 2011 Jul;118(1):29-38. doi: 10.1097/AOG.0b013e31821e5f65. PMID 21646928
- [Background] Carusi, D. A., & Goldberg, A. B. (2015). Intrauterine contraceptive device: insertion and removal. In: M. Zieman (Ed), UpToDate. Retrieved from http://www.uptodate.com/home .
- [Background] Centers for Disease Control and Prevention. (2013). U.S. selected practice recommendations for contraceptive use, 2013: Adapted from the World Health Organization selected practice recommendations for contraceptive use. Retrieved from http://www.cdc.gov/mmwr/pdf/rr/rr6205.pdf
- [Background] d'Arcangues C. Worldwide use of intrauterine devices for contraception. Contraception. 2007 Jun;75(6 Suppl):S2-7. doi: 10.1016/j.contraception.2006.12.024. Epub 2007 Apr 19. PMID 17531612
- [Background] Edmunds, M. W., & Mayhew, M. S. (2014). Pharmacology for the primary care provider (4th ed.). St. Louis, MI: Elsevier Mosby.
- [Background] Finer LB, Jerman J, Kavanaugh ML. Changes in use of long-acting contraceptive methods in the United States, 2007-2009. Fertil Steril. 2012 Oct;98(4):893-7. doi: 10.1016/j.fertnstert.2012.06.027. Epub 2012 Jul 13. PMID 22795639
- [Background] Fox MC, Krajewski CM. Cervical preparation for second-trimester surgical abortion prior to 20 weeks' gestation: SFP Guideline #2013-4. Contraception. 2014 Feb;89(2):75-84. doi: 10.1016/j.contraception.2013.11.001. Epub 2013 Nov 11. PMID 24331860
- [Background] Heikinheimo O, Inki P, Kunz M, Parmhed S, Anttila AM, Olsson SE, Hurskainen R, Gemzell-Danielsson K. Double-blind, randomized, placebo-controlled study on the effect of misoprostol on ease of consecutive insertion of the levonorgestrel-releasing intrauterine system. Contraception. 2010 Jun;81(6):481-6. doi: 10.1016/j.contraception.2010.01.020. Epub 2010 Mar 1. PMID 20472114
- [Background] Hubacher D, Reyes V, Lillo S, Zepeda A, Chen PL, Croxatto H. Pain from copper intrauterine device insertion: randomized trial of prophylactic ibuprofen. Am J Obstet Gynecol. 2006 Nov;195(5):1272-7. doi: 10.1016/j.ajog.2006.08.022. PMID 17074548
- [Background] Kass-Wolff JH, Fisher JE. Evidence-based pain management for endometrial biopsies and IUD insertions. Nurse Pract. 2014 Mar 13;39(3):43-50. doi: 10.1097/01.NPR.0000434094.19101.d1. PMID 24535311
- [Background] Lopez LM, Bernholc A, Zeng Y, Allen RH, Bartz D, O'Brien PA, Hubacher D. Interventions for pain with intrauterine device insertion. Cochrane Database Syst Rev. 2015 Jul 29;2015(7):CD007373. doi: 10.1002/14651858.CD007373.pub3. PMID 26222246
- [Background] Maguire K, Morrell K, Westhoff C, Davis A. Accuracy of providers' assessment of pain during intrauterine device insertion. Contraception. 2014 Jan;89(1):22-4. doi: 10.1016/j.contraception.2013.09.008. Epub 2013 Sep 21. PMID 24134898
- [Background] Singh RH, Thaxton L, Carr S, Leeman L, Schneider E, Espey E. A randomized controlled trial of nitrous oxide for intrauterine device insertion in nulliparous women. Int J Gynaecol Obstet. 2016 Nov;135(2):145-148. doi: 10.1016/j.ijgo.2016.04.014. Epub 2016 Jul 16. PMID 27481016
- [Background] Winner B, Peipert JF, Zhao Q, Buckel C, Madden T, Allsworth JE, Secura GM. Effectiveness of long-acting reversible contraception. N Engl J Med. 2012 May 24;366(21):1998-2007. doi: 10.1056/NEJMoa1110855. PMID 22621627
- [Background] Medical Eligibility Criteria for Contraceptive Use: A WHO Family Planning Cornerstone. 4th edition. Geneva: World Health Organization; 2010. Available from http://www.ncbi.nlm.nih.gov/books/NBK138639/ PMID 23741782
- [Background] Zhuo Z, Yu H, Jiang X. A systematic review and meta-analysis of randomized controlled trials on the effectiveness of cervical ripening with misoprostol administration before hysteroscopy. Int J Gynaecol Obstet. 2016 Mar;132(3):272-7. doi: 10.1016/j.ijgo.2015.07.039. Epub 2015 Dec 11. PMID 26797202